CLINICAL TRIAL: NCT01994148
Title: Study of Laparoscopy in Gastrointestinal Injury
Brief Title: Application of Laparoscopy in Gastrointestinal Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Zongguang Zhou (Other)
Responsible Party: Sponsor-Investigator, Prof. Zongguang Zhou, Director of gastrointestinal surgery center, WestChina Hospital, West China Hospital
Organization: West China Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LGI-201302016
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Gastrointestinal Injury
Keywords: Trauma; Gastrointestinal injury; Laparoscopy
MeSH Terms: conditions — Wounds and Injuries | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laparoscopy (Experimental): Laparoscopy has been increasingly applied in patients with abdominal trauma , as an diagnostic and therapeutic modality. In this arm, we will include 100 Hemodynamically stable patients with gastrointestinal trauma, all of them will receive laparoscopic exploration,laparoscopic repair of the gastrointestinal injury will be attempted.
  Interventions: Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Laparoscopy — In this study, laparoscopic intervention will be performed under carbon dioxide pneumoperitoneum (pressure, 10-12 mm Hg; flow volume, 8-10 L/min). A 12-mm trocar will be placed in the umbilicus with use of an open technique and to establish pneumoperitoneum.A 10-mm and a 5-mm trocar will be inserted in the right and left flanks,respectively.

SUMMARY:
laparoscopy has been increasingly applied in patients with abdominal trauma , as an diagnostic and therapeutic modality. However, its clinical benefits are still under evaluation. The aim of this study is to prospectively assess the feasibility and safety of this technique in the management of traumatic gastrointestinal injury.

DETAILED DESCRIPTION:
This prospective single arm study was undertaken in West China Hospital, Sichuan University, Chengdu, China. The institution is the largest medical center in southwest China, and also a national training center of laparoscopy. Surgeons participated in the study were well trained in gastrointestinal laparoscopy and hepatobiliary laparoscopy, and were experienced in management of abdominal trauma.

The study was approved by the institutional review committees. The participants provided written informed consent.

Patients age 18 years or older with abdominal trauma were considered eligible, regardless of the nature of trauma (blunt or penetrating), but hemodynamic stability was mandatory.

Patients meet the following criteria is prepared for laparoscopic exploration:

Evidence showed that wound penetrates the peritoneum in penetrating trauma or/and signs of peritoneal irritation or positive CT scan in those without penetration of peritoneum and patients with blunt injuries.

We defined the CT scan positive by it shows peritoneal effusion, free intraperitoneal air, fat density increase, substantive organ rupture and intestinal wall swelling and other signs of abdominal trauma.

Laparoscopic screening will be performed according to protocol. The study demands that all surgeons should complete the repair laparoscopically as much as possible when condition allow, and record reasons for conversion in detail when it is inevitable.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gastrointestinal trauma
* Blood loss < 1000ml
* Hemodynamically stable
* Vital sign is stable
* Willing to comply to the study procedure and complete the study.

Exclusion Criteria:

* Severe hemorrhage or intraperitoneal infections
* Combined with other conditions which are contraindications to laparoscopy
* Pregnant or lactating woman
* Severe immunodeficiency
* History of drug abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 3 month after operation

SECONDARY OUTCOMES:
Number of iatrogenic injury during the operation | at the end of the operation
Number of patients with postoperative complications | up to 3 months
  Postoperative complications include bowel obstruction, wound infection, postoperative hemorrhage,intestine fistula
Operative time | at the end of the operaion
Blood loss during the operation | at the end of the operation
Length of hospital stay | 1 month
Number of patients transferred to open operation | at the end of the operation

CONTACTS AND LOCATIONS:
Overall Officials: Zongguang Zhou, MD., PhD, Study Chair — West China Hospital
Locations (4):
- China (4):
  - Xijing Hospital, The 4th Militory Medical University, Xian, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Chinese PLS General Hospital, Beijing
  - Southwest Hospital, The 3rd Militory Medical University, Chongqing